CLINICAL TRIAL: NCT04526873
Title: Encouraging Annual Wellness Visits Among Keystone ACO Beneficiaries
Brief Title: Encouraging Annual Wellness Visits Among ACO Beneficiaries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Amir Goren, Program Director, Behavioral Insights Team, Geisinger Clinic
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2020-0577
Record Dates: First submitted 2020-08-14; First posted 2020-08-26 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Health Promotion; Prevention; Risk Reduction Behavior; Telehealth
Keywords: Behavioral Economics; Humor; Salience; Present Bias
MeSH Terms: conditions — Risk Reduction Behavior | interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: Postcard content will follow a factorial design (crossing telehealth vs. non-telehealth with cartoon/salience vs. stock photo). In addition, there will be a no-contact control group and a phone call group.
Who Masked: Participant, Care Provider
Masking Description: Participants (i.e., patients) will not be informed specifically of their assignment to different arms throughout the study. Providers who conduct AWVs will not be randomized to study arms or informed of patient assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Control (No Intervention): No intervention control group
- Postcard: non-telehealth, photo (Experimental): This group receives a postcard that does not include telehealth information and features a stock photo
  Interventions: Behavioral: Postcard
- Postcard: non-telehealth, salience/humorous cartoon (Experimental): This group receives a postcard that does not include telehealth information and features a humorous cartoon as well as examples of serious health risks that the visit could help prevent (stroke and heart attack)
  Interventions: Behavioral: Postcard; Behavioral: Humor/Salience
- Postcard: telehealth, photo (Experimental): This group receives a postcard that does includes telehealth information and features a stock photo
  Interventions: Behavioral: Postcard; Behavioral: Telehealth
- Postcard: telehealth, salience/humorous cartoon (Experimental): This group receives a postcard that includes telehealth information and features a humorous cartoon as well as examples of serious health risks that the visit could help prevent (stroke and heart attack)
  Interventions: Behavioral: Postcard; Behavioral: Humor/Salience; Behavioral: Telehealth
- Phone call (Experimental): This group receives a phone call
  Interventions: Behavioral: Phone call

INTERVENTIONS:
Behavioral: Postcard — Mailed
  Arms: Postcard: non-telehealth, photo; Postcard: non-telehealth, salience/humorous cartoon; Postcard: telehealth, photo; Postcard: telehealth, salience/humorous cartoon
Behavioral: Phone call — May be automated or by human
  Arms: Phone call
Behavioral: Humor/Salience — Funny cartoon + health risk examples
  Arms: Postcard: non-telehealth, salience/humorous cartoon; Postcard: telehealth, salience/humorous cartoon
Behavioral: Telehealth — Information about video visit
  Arms: Postcard: telehealth, photo; Postcard: telehealth, salience/humorous cartoon

SUMMARY:
Annual Wellness Visits (AWVs) are a type of detailed healthcare checkup to which Medicare beneficiaries are entitled, free of charge, once per year. The purpose of the current study is to assess what content and communication modality results in the most effective messaging campaign to encourage Medicare beneficiaries to schedule their AWVs.

DETAILED DESCRIPTION:
Annual Wellness Visits (AWVs) are a type of detailed healthcare checkup to which Medicare beneficiaries are entitled, free of charge, once per year. The Keystone Affordable Care Organization (KACO), of which Geisinger is a part, is working to increase the number of eligible patients who take advantage of AWVs via mail and telephone outreach.

The purpose of the current study is to assess what content and communication modality results in the most effective messaging campaign. Patients will either receive a phone call or a mailed postcard, or they will be part of a no-contact control condition. Furthermore, the content of the postcard will vary in terms of humor and salience, as well as whether telehealth is mentioned as an AWV option.* Although telehealth is a great option for patients who are unable to attend an in-person visit, the latter is preferable in terms of quality of care. Furthermore, insurance coverage for telehealth visits may not extend indefinitely beyond the COVID-19 pandemic. Highlighting the telehealth option may help attract patients who would not otherwise get an AWV, increasing the effectiveness of the intervention. On the other hand, it may unintentionally nudge patients who would otherwise have scheduled an in-person visit to opt for telehealth instead.

The following research questions will assess effectiveness in increasing patient scheduling of an AWV:

1. Are postcards effective compared with a no-contact control condition?
2. How effective are postcards when compared with phone calls, a presumably more intrusive type of intervention?
3. Is a humorous cartoon, accompanied by language using examples to make salient the future health risks that could be prevented, more effective than stock photography of similar patient-doctor situations (typically used in outreach), accompanied by prevention language that is less specific?
4. Is it more effective to highlight the availability of telehealth video visits than not to mention that option?
5. Are in-person AWVs are scheduled at least as frequently when the telehealth option is highlighted as when it is not?

Included in the study will be patients from 7 KACO partner sites: Caring Community Health Center, Evangelical Community Hospital, Geisinger, Geisinger-Hm Joint Venture, Holy Spirit, Wayne Memorial Hospital, and Wright Center. Generalized linear mixed models (GLMMs) will examine the primary study outcomes as a function of the study arms (between-subjects), with partner site included as a random effect, assuming high intraclass correlation coefficients.

* Wayne Memorial Hospital patients will not receive postcards with tele-health content. In addition, only patients from the following partner sites will be randomized to receive a phone call: Evangelical Community Hospital, Wayne Memorial Hospital, and the Wright Center. Geisinger patients will not be randomized to receive phone calls, but Geisinger patients who are randomized to other conditions may receive phone calls as part of regular operations. This will be accounted for during analysis as a model regressor.

ELIGIBILITY:
Inclusion Criteria:

* KACO Medicare beneficiary
* Haven't had an AWV or due for their next one
* For phone call condition only: patients of Evangelical Community Hospital, Wayne Memorial Hospital, and the Wright Center

Exclusion Criteria:

* Patient has already been called about AWV or had a visit scheduled
* For "patient initiated contact" outcome only: patients of Wayne Memorial Hospital or who have not been assigned to a partner site. This is because postcards received by these patients will not include a specific phone number to call.
* For telehealth conditions only: patients of Wayne Memorial Hospital

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41472 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who scheduled an AWV appointment | 1 month after start of intervention
  Patient scheduled an AWV appointment
Proportion of patients who completed an AWV visit | 3 months after start of intervention
  Patient completed an AWV

SECONDARY OUTCOMES:
Proportion of patients who scheduled an AWV appointment | 3 months after start of intervention
  Patient scheduled an AWV appointment
Proportion of patients who initiated contact | 3 months after start of intervention
  Patient called one of the phone numbers provided on postcards regarding AWV
Proportion of visits that were in-person vs. tele-visit | 3 months after start of intervention
  Whether patient AWV was in person or a telehealth visit

OTHER OUTCOMES:
Per patient campaign cost | 3 months after start of intervention
  Cost of campaign for whole study arm divided by number of patients who completed an AWV for that study arm.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Goren, PhD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No